CLINICAL TRIAL: NCT00373230
Title: Treating Obesity and Its Consequences in Underserved Overweight Populations
Brief Title: Treating Obesity in Underserved Overweight Populations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Temple University (Other)
Collaborators: Geisinger Clinic (Other); University of Pennsylvania (Other); Insight Telehealth Systems (Industry)
Responsible Party: Guenther Boden, MD, Temple University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005NFGrantTemple
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Overweight
Keywords: weight loss; telemedicine; african-american; rural
MeSH Terms: conditions — Overweight; Weight Loss | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Internet based telemedicine weight maintenance program
  Interventions: Behavioral: telemedicine
- 2 (Active Comparator): In person weight maintenance monthly consultations
  Interventions: Behavioral: telemedicine

INTERVENTIONS:
Behavioral: telemedicine — One year behavioral modification weight control program comparing in-person consultations (monthly) to a computer based telemedicine system (available 24/7).

SUMMARY:
Obesity has reached epidemic proportions with nearly two-thirds of the US population either overweight or obese. Thus, novel strategies that both improve weight loss maintenance and are accessible to those most in need are the focus of this application, which will determine if a telemedicine system can help participants, who have undergone a weight loss program based in church and community centers, maintain their weight loss over a 1 year period. Telemedicine will provide support through self-monitoring, education, supervised chat room, bulletin board, and e-mail.

DETAILED DESCRIPTION:
Obesity has reached epidemic proportions with nearly two-thirds of the US population either overweight or obese. Ethnic minorities are disproportionately affected with 37% of African-American adults being obese. Obesity is also inversely related to socioeconomic status. In Pennsylvania, the prevalence of obesity increased from 14.7% in 1991 to 24.0% in 2002, and annual medical expenditures attributable to obesity are estimated at $4.2 billion; making Pennsylvania the 4th highest state in the country in terms of obesity-related costs. The prevalence of obesity is matched by it serious medical consequences including type 2 diabetes, hypertension, dyslipidemia, and atherosclerotic disease. The core pathogenetic factor underlying these conditions appears to be insulin resistance. Weight loss through diet and physical activity is the most desirable way to reduce insulin resistance (IR). Weight losses of 8-10% are associated with significant improvements in IR. While clinic-based weight loss programs at tertiary medical centers can produce clinically significant losses, the cost and location of these programs make them inaccessible to underserved populations (e.g., inner city African Americans and rural poor) who are most in need. Moreover, the most common outcome for weight loss treatments is weight regain. Thus, novel strategies that both improve weight loss maintenance and are accessible to those most in need are a priority for research and the focus of this application.

Based on our expertise in behavioral weight management and telemedicine, this study will determine if a telemedicine system can help participants, who have undergone a weight loss program based in church and community centers, maintain their weight loss over a 1 year period. Overweight and obese men and women (n = 400) will participate in a 16-week behavioral weight loss program in local churches and community centers. After 16 weeks, participants will be randomized to either an "In-person" follow-up group or to a "telemedicine" group for 1-year. The latter will provide support through self-monitoring, education, supervised chat room, bulletin board, and e-mail. Assessments of body weight, body composition and insulin sensitivity will be conducted at baseline, 16 and 68 weeks. Based on recent data, we predict greater maintenance of weight loss (and lower body weights) at 68 weeks in the Telemedicine group as compared to the "In person group".

ELIGIBILITY:
Inclusion Criteria:

* 27<BMI<45
* Able to walk

Exclusion Criteria:

* Diabetes on medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-02 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
subject's weight | 3 and 15 months

SECONDARY OUTCOMES:
Use of telemedicine system | over 12 months
blood lipids | 3 and 15 months
blood glucose | 3 and 15 months
A1c | 3 and 15 months
Insulin | 3 and 15 months
blood pressure | 3 and 15 months
Oral Glucose Tolerance | 3 and 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Boden, MD, Principal Investigator — Temple University
Locations (2):
- United States (2):
  - Geisinger Medical Center, Danville, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania